CLINICAL TRIAL: NCT00816660
Title: Recombinant Von Willebrand Factor / Recombinant Factor VIII Complex (rVWF:rFVIII): A Phase 1 Study Evaluating the Pharmacokinetics (PK), Safety, and Tolerability in Type 3 Von Willebrand Disease (VWD)
Brief Title: Pharmacokinetic, Safety and Tolerability Study of Recombinant Von Willebrand Factor / Recombinant Factor VIII Complex in Type 3 Von Willebrand Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baxalta now part of Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 070701
Record Dates: First submitted 2009-01-02; First posted 2009-01-05 (Estimated); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Von Willebrand Disease
MeSH Terms: conditions — von Willebrand Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Biological: Recombinant von Willebrand factor : recombinant FVIII (rVWF:rFVIII)
- 2 (Active Comparator)
  Interventions: Biological: Recombinant von Willebrand factor : recombinant FVIII (rVWF:rFVIII); Biological: Marketed plasma-derived VWF/FVIII concentrate

INTERVENTIONS:
Biological: Recombinant von Willebrand factor : recombinant FVIII (rVWF:rFVIII) — Single dose, dose escalation, various cohorts
Biological: Marketed plasma-derived VWF/FVIII concentrate — Cross-over: recombinant FVIII (rVWF:rFVIII) and marketed plasma-derived VWF/FVIII concentrate
  Arms: 2

SUMMARY:
The objectives of this study are to evaluate the immediate tolerability and safety of rVWF:rFVIII in subjects with Type 3 Von Willebrand Disease after administration of various dosages of VWF:RCo.

ELIGIBILITY:
Inclusion Criteria:

* Subject has voluntarily given written informed consent (before conduct of any study-related procedures)
* The subject has hereditary type 3 VWD (<= 3 IU/dL VWF:Ag)or severe type 1 or type 2A VWD (VWF:RCo <= 10% and FVIII:C <20%)
* The subject has a medical history of at least 25 exposure days to VWF/FVIII coagulation factor concentrates
* The subject has a Karnofsky score >= 70%
* The subject is between 18 to 60 years of age (on the day of signing the informed consent)
* NOT APPLICABLE IN ITALY: Female subjects of child-bearing potential must have a negative pregnancy test and agree to practice contraception using a method of proven reliability from the day of screening until the study completion visit
* APPLICABLE ONLY IN ITALY: Female subjects of child-bearing potential must have a negative pregnancy test and agree to practice non-hormonal-based contraception using a method of proven reliability (IUD acceptable) from the day of screening until 96 hours after the last investigational drug infusion
* NOT APPLICABLE IN ITALY: The subject must agree not to be on any therapy (hormone-based contraception acceptable) interfering with coagulation factor pharmacokinetics until 96 hours after the last investigational drug infusion
* APPLICABLE ONLY IN ITALY: The subject must agree not to be on any therapy interfering with coagulation factor pharmacokinetics until 96 hours after the last investigational drug infusion

Exclusion Criteria:

* The subject has been diagnosed with a hereditary or acquired coagulation disorder other than VWD (including qualitative and quantitative platelet disorders and/or an international normalized ratio (INR) > 1.4)
* The subject has been diagnosed with an ADAMTS13 deficiency with less than 10% ADAMTS13 activity
* The subject has a history or presence of VWF inhibitor
* The subject has a history or presence of FVIII inhibitor with a titer >= 0.4 BU (by Nijmegen assay) or >= 0.6 BU (by Bethesda assay)
* The subject has a known hypersensitivity to mouse or hamster proteins
* The subject has a medical history of immunological disorders, excluding seasonal allergic rhinitis/conjunctivitis, food allergies or animal allergies
* The subject has a medical history of a thromboembolic event
* The subject is HIV positive with an absolute CD4 count < 200/mm3
* The subject has been diagnosed with cardiovascular disease (New York Heart Association (NYHA) classes 1-4)
* The subject has been diagnosed with insulin-dependent diabetes mellitus
* The subject has an acute illness (e.g. influenza, flu-like syndrome, allergic rhinitis/conjunctivitis)
* The subject has been diagnosed with liver disease, as evidenced by, but not limited to, any of the following: serum ALT three times the upper limit of normal, hypoalbuminemia, portal vein hypertension (e.g. presence of otherwise unexplained splenomegaly, history of esophageal varices)
* The subject has been diagnosed with renal disease, with a serum creatinine level >= 2 mg/dL
* In the judgment of the investigator, the subject has another clinically significant concomitant disease (e.g. uncontrolled hypertension, diabetes type II) that may pose additional risks for the subject
* The subject has been treated with an immunomodulatory drug, excluding topical treatment (e.g. ointments, nasal sprays) within 30 days before enrollment
* The subject has been treated with drugs known to induce thrombotic thrombocytopenic purpura (TTP) (e.g. Adenosine diphosphate (ADP) receptor inhibitors (Clopidogrel, Ticlopidine)) within 60 days before enrollment
* The subject is receiving or anticipates receiving another investigational and/or interventional drug within 30 days before enrollment
* The subject is a lactating female
* The subject has a history of drug or alcohol abuse within the last 5 years
* The subject has a progressive fatal disease and/or life expectancy of less than 3 months
* The subject is identified by the investigator as being unable or unwilling to cooperate with study procedures
* The subject suffers from a mental condition rendering him/her unable to understand the nature, scope and possible consequences of the study and/or evidence of an uncooperative attitude
* Subject is in prison or compulsory detention by regulatory and/or juridical order

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2008-12-01 (Actual); Primary Completion 2010-08-31 (Actual); Study Completion 2010-08-31 (Actual)

PRIMARY OUTCOMES:
To demonstrate the immediate tolerability and safety after single-dose injections of rVWF:rFVIII at various doses | Up to 30 days after the last investigational product infusion

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (25):
- United States (10):
  - Emory University School of Medicine, Dept. of Pediatrics, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Indiana Hemophilia and Thrombosis Center, Indianapolis, Indiana
  - University of Kentucky Hemophilia Treatment Center, Lexington, Kentucky
  - Brown Cancer Center, Louisville, Kentucky
  - Brigham & Women´s Hospital, Hematology Division, Boston, Massachusetts
  - Rochester General Hospital, Rochester, New York
  - Hemophilia Center of Western PA, Pittsburgh, Pennsylvania
  - University of Texas, Houston, Texas
  - Comprehensive Center for Bleeding Disorders, Milwaukee, Wisconsin
- General Hospital Vienna (Allgemeines Krankenhaus der Stadt Wien), University Department for Internal Medicine I, Vienna, Austria
- Q.E.II Health Sciences Centre, Halifax, Nova Scotia, Canada
- Germany (3):
  - Vivantes Klinikum im Friedrichshain, Berlin
  - Hannover Medical School - Clinic for Haematology, Haemostaseology, Oncology and Stem Cell Transplantation, Hanover
  - Institut für Thrombophilie und Hämostaseologie, Münster
- Italy (6):
  - Azienda Ospedaliero-universitaria "Careggi", Florence
  - Giannia Gaslini Children´s Hospital, Genova
  - Ospedale Maggiore di Milano, Centro Emofilia e Trombosi "Angelo Bianchi Bonomi", Milan
  - Ospedale San Giovanni Bosco, Centro Emofilia Divisione di Ematologia, Naples
  - University of Padua Medical School, Padua
  - Ospedale di Vicenza - U.L.S.S.N.6, Vicenza
- United Kingdom (4):
  - West Midlands Region Adult Haemophilia Centre, Queen Elizabeth Hospital, Birmingham
  - Imperial College School of Medicine, Hammersmith Hospital, London
  - Central Manchester Healthcare NHS Trust, Manchester Haemophilia Comprehensive Care Centre, Manchester
  - Royal Cornwall Hospital, Truro

REFERENCES:
- [Derived] Mannucci PM, Kempton C, Millar C, Romond E, Shapiro A, Birschmann I, Ragni MV, Gill JC, Yee TT, Klamroth R, Wong WY, Chapman M, Engl W, Turecek PL, Suiter TM, Ewenstein BM; rVWF Ad Hoc Study Group. Pharmacokinetics and safety of a novel recombinant human von Willebrand factor manufactured with a plasma-free method: a prospective clinical trial. Blood. 2013 Aug 1;122(5):648-57. doi: 10.1182/blood-2013-01-479527. Epub 2013 Jun 18. PMID 23777763